CLINICAL TRIAL: NCT05434299
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of TFX05-01 in Participants With Advanced Malignancies
Brief Title: A Study of TFX05-01 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Yangli Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-TFX05-01-2021-C001
Record Dates: First submitted 2022-06-10; First posted 2022-06-28 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Single agent dose escalation
  Interventions: Drug: TFX05-01
- Dose expansion (Experimental): Single agent dose expansion
  Interventions: Drug: TFX05-01

INTERVENTIONS:
Drug: TFX05-01 — TFX05-01 for intravenous

SUMMARY:
This is an open-label, non-randomized, multicenter, Phase Ⅰ/Ⅱa study to evaluate the safety, tolerability, pharmacokinetics and efficacy of TFX05-01 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study to evaluate the safety, tolerability, pharmacokinetics and efficacy of TFX05-01 in patients with advanced solid tumors, which was divided into dose exploration part (Phase Ⅰ) and indication exploration part (Phase Ⅱa). Each Phase of the study consisted of a screening period (21 days before initial dosing), a treatment period (from the first trial to the onset of an endpoint event), and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 18 years of age at the time of screening. And participants ≤75 years of age for phase Ⅰ.
* All toxicities from prior therapy (except for alopecia, fatigue, or peripheral neuropathy) must have returned to grade 0 or 1 (NCI CTCAE 5th edition) before initiation of the study drug.
* Subjects with advanced malignant solid tumors confirmed by histopathology/cytology or clinical diagnosis, who are not suitable for surgery or local therapy, or whose disease has progressed after surgery and/or last-line standard therapy and/or cannot tolerate standard therapy.
* Subjects have at least one measurable lesion that meets RECIST 1.1 criteria. Lesions previously irradiated are not considered measurable lesions unless they show clear radiographic progression after radiotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Life expectancy ≥ 12 weeks.
* The cardiac QTcF interval is ≤ 450 ms in males and ≤ 470 ms in females.
* Laboratory tests must meet the following criteria:

  1. Hematologic function (no blood transfusion or cell growth factor correction within 14 days before screening): hemoglobin ≥ 90 g/L, platelet count ≥ 100 × 10^9/L, absolute neutrophil count (ANC) ≥1.5 × 10^9/L;
  2. Hepatic and renal function (no albumin infusion within 14 days before screening): creatinine clearance >60 mL/min measured by Cockcroft-Gault equation. Serum total bilirubin ≤2.5 times the upper limit of normal (ULN); ALT and AST≤2.5 × ULN (AST and ALT ≤5×ULN for patients with comorbidities liver metastases);
  3. Coagulation function: International normalized ratio (INR) ≤2.3 or activated partial prothrombin time (APTT) < 1.5 times the upper limit of normal.
* No history of alcohol, drug, or substance abuse in the past year.
* Female subjects of childbearing potential must be non-lactation and have a negative serum pregnancy test performed within 7 days before the start of treatment. Infertile female subjects must meet at least one of the following criteria:

  1. Postmenopausal status, defined as follows: cessation of regular menstruation for at least 12 consecutive months, with no other pathological or physiological cause; serum follicle-stimulating hormone (FSH) level confirmed postmenopausal status;
  2. Had undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Medically confirmed ovarian failure;
  4. All other female subjects (including those with tubal ligation) were considered fertile.
* Female and male subjects of reproductive potential must agree to use effective contraception with their partner (e.g. surgical sterilization or condom or diaphragm contraception combined with spermicidal gel or intrauterine device) from study participation until 3 months after the last dose of the study drug.
* Subjects must voluntarily participate in the study and fully understand the risks, have good compliance, and sign informed consent.

Exclusion Criteria:

* Untreated active central nervous system (CNS) metastases, brain metastases, or leptomeningeal disease. Subjects may participate in the study if their CNS metastases had been adequately treated and were stable for at least 4 weeks as confirmed by clinical examination and brain imaging (MRI or CT) during screening.
* More than 25% of the bone marrow had previously received radiotherapy.
* Have a history of severe allergies in the past, or are allergic to any active or inactive ingredients (phosphates, etc.) of the study drug.
* Major surgery other than diagnostic surgery within 4 weeks before the first dose of the study drug.
* Subjects who received radiation therapy, surgery, chemotherapy, immunotherapy, biological therapy for cancer, targeted therapy, or hormonal therapy within 4 weeks before the first dose of the study drug (exceptions: nitrosourea or mitomycin C therapy needs a 6-week washout period; oral fluorouracil, requiring a 2-week washout period; small molecule targeted therapy demands a 2-week washout period).
* Bleeding tendency and history of thrombosis: (1) Clinically significant bleeding symptoms or clear bleeding tendency within 3 months before screening; (2) History of gastrointestinal bleeding or clear gastrointestinal bleeding tendency within 6 months before screening; (3) Arterial/venous thrombotic events, such as cerebrovascular accident (including transient ischemic attack), within 6 months before screening.
* History of severe cardiovascular disease : (1) NYHA (New York Heart Association) grade 3 and 4 congestive heart failure; (2) unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening; (3) CTCAE ≥ grade 2 valvular heart disease; (4) hypertension (systolic blood pressure>150mmHg or diastolic blood pressure>90mmHg) poorly controlled by drugs.
* Subjects have any active, known, or suspected autoimmune disease.
* Clinically significant ascites, defined as detected by physical examination and requiring control by abdominocentesis, or increased medical intervention to maintain symptoms (patients with ascites detected only by imaging were eligible).
* Participated in a drug study (diagnostic or therapeutic) or device study within 4 weeks before the first dose of the study drug.
* A combination of potent inhibitors or inducers of CYP3A and CYP2C8 was required during the study.
* An active bacterial, viral or fungal infection that has not been controlled and requires systemic treatment.
* Known infection with human immunodeficiency virus (HIV) or positive for syphilis.
* Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Concomitant diseases or symptoms that may interfere with the conduct of the study, or physical abnormalities that the investigator considers posing an excessive risk to the subjects, including but not limited to active peptic ulcer or gastritis, changes in mental status, or mental abnormalities that may interfere with the subject's understanding of informed consent.
* Subjects who are unwilling or unable to comply with the study protocol for any reason.
* Subjects who are judged by the investigator to be unsuitable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AE) [Safety and Tolerability] | Through study completion (About two years)
  AE will be graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Electrocardiogram (ECG) changes [Safety and Tolerability] | Through study completion (About two years)
  Resting 12-lead ECGs will be obtained from all subjects in order to assess any impact TFX05-01 may have on the QT interval as assessed by the Fridericia's Correction Formula (QTcF).
Monitoring of Vital signs [Safety and Tolerability] | Through study completion (About two years)
  Vital sign will be obtained from all subjects.
Monitoring of hematology and blood chemistry [Safety and Tolerability] | Through study completion (About two years)
  Hematology and blood chemistry will be obtained from all subjects.
Monitoring of coagulation function [Safety and Tolerability] | Through study completion (About two years)
  Coagulation function will be obtained from all subjects.
Monitoring of urinalysis [Safety and Tolerability] | Through study completion (About two years)
  Urinalysis will be obtained from all subjects.
Maximum tolerated dose (MTD) | Through the end of the first cycle (Days 1-21)
  MTD as determined by percentage of participants with dose limiting toxicities (DLTs).
Recommended Phase 2 Dose (RP2D) | Through study completion (About two years)
  RP2D as determined by percentage of participants with DLTs and cumulative safety.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) - Time to maximum concentration (Tmax) | Throughout Days 1 and 8 of Cycle 1 and Days 1 of Cycle 2-N (21 days for each cycle)
  Tmax of TFX05-01 will be computed for each subject where possible.
PK - Maximum peak plasma concentration (Cmax) | Throughout Days 1 and 8 of Cycle 1 and Days 1 of Cycle 2-N (21 days for each cycle)
  Cmax of TFX05-01 will be computed for each subject where possible.
PK - Terminal Elimination Half-life (T1/2) | Throughout Days 1 and 8 of Cycle 1 and Days 1 of Cycle 2-N (21 days for each cycle)
  T1/2 of TFX05-01 will be computed for each subject where possible.
PK -Area under the plasma concentration versus time curve (AUC) | Throughout Days 1 and 8 of Cycle 1 and Days 1 of Cycle 2-N (21 days for each cycle)
  AUC of TFX05-01 will be computed for each subject where possible.
The overall response rate (ORR) | Through study completion (About two years)
  ORR will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1.
Duration of response (DoR) | Through study completion (About two years)
  DoR assessed by RECIST 1.1 criteria.
Disease control rate (DCR) | Through study completion (About two years)
  DCR assessed by RECIST 1.1 criteria.
Progression free survival (PFS) | Through study completion (About two years)
  PFS assessed by RECIST 1.1 criteria.
Overall survival (OS) | Through study completion (About two years)
  The time from randomization to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences，study principal investigator
Locations (4):
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The 1st Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No